CLINICAL TRIAL: NCT05800717
Title: A Self-Management Program for Improving the Well-Being of Veterans With AIS D Incomplete Spinal Cord Injury
Brief Title: Self-Management Program for AIS D SCI
Acronym: SCISM-D
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4417-P; 1I21RX004417-01A1 (NIH)
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Psychological Well-Being; Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Psychological Well-Being; Clinical trial
MeSH Terms: conditions — Psychological Well-Being; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: single group, successive cohort design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): Receives SCISM-D.
  Interventions: Behavioral: SCI Self-Management for AIS D

INTERVENTIONS:
Behavioral: SCI Self-Management for AIS D — An individually administered, self-management intervention for Veterans with AIS D spinal cord injury.

SUMMARY:
About 25-51% of adults with acquired spinal cord injury (SCI) have "AIS D" SCI, the lowest severity grade of neurologic injury. Veterans with AIS D SCI generally have better outcomes in mobility, community integration, and employment. However, counterintuitively, they are also at higher risk of poor subjective well-being (SWB) and related psychosocial outcomes. Preliminary evidence suggests that poorer SWB in this group is associated with distinctive, modifiable factors such as less intensity of acute rehabilitation services, limited development of instrumental and social support networks, and underdeveloped disability identity. A significant gap in the care of Veterans with AIS D SCI is that they are unlikely to receive rehabilitation that is responsive to their specific experiences and needs. The proposed study will develop a novel, self-management based program to help Veterans with AIS D SCI. This study is highly significant, as creation of the proposed program is expected to improve SWB and lifetime psychosocial functioning for Veterans with AIS D SCI.

DETAILED DESCRIPTION:
Background and Significance: Spinal cord injury (SCI) is a life-altering event that often results in permanent paralysis and sensory loss, with subsequent loss of physical function and independence and risk for negative psychosocial outcomes. About 25-51% of adults with acquired SCI have AIS D SCI and have an excellent prognosis for ambulation, are less visibly disabled, and generally have better objective well-being, such as community integration and mobility. However, counterintuitively, military Veterans with AIS D SCI are at higher risk of poor subjective well-being (SWB) including higher rates of depression and suicidal ideation. Several factors that may explain the disparity in well-being have been proposed, including less acute rehabilitation services, limited development of instrumental and social support networks, greater prevalence of comorbid health issues, and underdeveloped disability identity. Given that SWB is central to quality of life, it is essential to understand and foster those skills, perspectives, and resources that best support SWB after SCI.

Specific Aims: This study will develop the first intervention targeting the well-being of Veterans with AIS D SCI by attending to their specific needs using a self-management approach. Self-management (SM) programs are differentiated by fostering engagement, knowledge, and authority to direct care to the patient. An SM-oriented program that is tailored to the needs and treatment preferences of Veterans with AIS D SCI has great promise to improve well-being. For this reason, the proposed study will develop the SCI Self- Management for AIS D (SCISM-D) Program, an individually administered, personalized support and skills training intervention via the VA's video telehealth-to-home technology, to improve well-being among Veterans with AIS D SCI. This study is highly significant for Veteran health care, as creation of the proposed SCISM-D program is expected to fill a critical health care gap and improve lifetime psychosocial functioning for Veterans with AIS D SCI. This study has three aims: (Aim 1) Develop SCISM-D to enhance the SWB of military Veterans with AIS D SCI using preliminary research and focus groups. (Aim 2) Conduct a pilot study to improve SCISM-D and test the feasibility and acceptability of SCISM-D to prepare for a future randomized controlled trial. (Aim 3) Finalize the SCISM-D program manual and consumer handbook.

Research Plan: For Aim 1, two focus groups of 4-6 Veterans with AIS D SCI and two focus groups of 4-6 SCI providers will be recruited to review, rate, and discuss proposed components of SCISM-D during two meetings each. Informed by the focus group ratings and feedback, the SCISM-D program manual and consumer handbook will be developed. Individual program components will be adapted from extant SM manuals with others developed by the investigators. The completed program manual and consumer handbook will then be presented to the focus groups and expert panel for feedback, followed by a final round of revisions. Criteria for success include completion of the focus groups and materials according to the study timeline.

Next, a pilot study will be conducted to examine the feasibility of SCISM-D and a subsequent randomized controlled trial (Aim 2). A target of 20 Veterans with AIS D SCI will complete the study. SCISM-D is anticipated to involve 5-7, 45-60-minute sessions conducted via the VA's telehealth system. Several measures and interviews will be administered during the program to assess treatment gains and mediators. Criteria for success include the ability to recruit at least 2 participants per month, at least 75% retention, at least 75% patient satisfaction, and an average change of "minimally improved" in confidence and life satisfaction, among others. After the pilot study, the focus group members will be asked to review the draft SCISM-D program manual and consumer handbook to inform final revisions to content by the team of investigators and layout by professional designers (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. VA clinician-confirmed diagnosis of tetraplegia or paraplegia with an ASIA rating of AIS D [Veterans with AIS D SCI];
2. Interest and ability (e.g., reliable video telehealth equipment and WiFi) to participate in the focus groups.

Exclusion Criteria:

1. Currently participating in a comprehensive, inpatient rehabilitation program;
2. Diagnosis of a psychotic disorder;
3. At high risk for suicidal/homicidal behavior;
4. Active substance dependence;
5. Lack of capacity to consent to participation;
6. Any medical condition that could affect results such as advanced cancer or neurologic disease such as Parkinson's disease; and
7. Mental disorders such as posttraumatic stress disorder and depressive disorder will not be exclusions, but any medications must have been stable for at least 30 days prior to enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 6 weeks
  An 8-item measure of patient satisfaction with the intervention. Each item is rated on a 4-point scale. The full scale has a range of 8-32 with higher scores indicating more satisfaction.
Patient Global Impression of Change | 6 weeks
  A one-item measure of self-reported change as a result of the intervention. Each item is rated on a 7-point scale: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: Scott D McDonald, PhD, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No